CLINICAL TRIAL: NCT06241833
Title: Effects of PPI on GI Bleeding and Cardiovascular Outcomes Among Post-MI Patients Taking DAPT
Brief Title: Emulation of Randomized Clinical Trial in Cardiovascular Disease
Acronym: RCT-BigData
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ki Hong Choi, Professor, Samsung Medical Center
Other Study IDs: CVD-Emulation
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
Keywords: Percutaneous coronary intervention; Cardiovascular Pharmacotherapy; Proton pump inhibitor; Dual antiplatelet therapy
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PPI group: Patients receiving PPI concomitant with dual antiplatelet therapy after PCI for AMI
  Interventions: Drug: PPI
- no PPI group: Patients receiving dual antiplatelet therapy only after PCI for AMI

INTERVENTIONS:
Drug: PPI — use of PPI concomitant with DAPT
  Other Names: GI protection
  Groups: PPI group

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study from Korean National Health Insurance Service database. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice.

ELIGIBILITY:
Inclusion Criteria:

* - PCI with MI (I21) admission
* Age more than 40 or less than 80 years old
* Aspirin and Clopidogrel/Prasugrel/Ticagrelor prescription with more than 2 days at discharge

Exclusion Criteria:

* - Previous use of a PPI, an H2-receptor antagonist, sucralfate, or misoprostol within 30 days before admission
* Preexisting cancer within a year before admission
* History of RBC transfusion
* RBC transfusion in admission
* Cardiogenic Shock
* Length of stay more than 14 days
* OAC prescription with more than 2 days at discharge
* H2 prescription with more than 2 days at discharge

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AMI undergoing PCI
Sampling Method: Non-Probability Sample
Enrollment: 118420 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of Major GI bleeding requiring transfusion | 1-year follow-up
  Efficacy outcome
Rates of Major adverse cardiac event | 1-year follow-up
  Safety outcome, a composite of cardiac death, MI, ischemic stroke, and repeat revascularization

SECONDARY OUTCOMES:
Rates of Major or Minor GI bleeding with hospitalization | 1-year follow-up
  Efficacy outcome
Rates of Cardiac death | 1-year follow-up
  Cardiac death
Rates of Spontaneous MI | 1-year follow-up
  Spontaneous MI
Rates of Ischemic stroke | 1-year follow-up
  Ischemic stroke
Rates of Repeat revascularization | 1-year follow-up
  Repeat revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Ki Hong Choi, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang D, Choi KH, Park H, Heo J, Park TK, Lee JM, Cho J, Yang JH, Song YB, Choi SH, Gwon HC, Hahn JY. Effects of proton pump inhibitors on gastrointestinal bleeding and cardiovascular outcomes in myocardial infarction patients treated with DAPT. EuroIntervention. 2025 Feb 17;21(4):e229-e239. doi: 10.4244/EIJ-D-24-00673. PMID 39962947